CLINICAL TRIAL: NCT01217151
Title: Perioperative Hemodynamic Goal-directed Optimization Using the Noninvasive NICOM™ Monitoring Device in Major Abdominal Surgery
Brief Title: Perioperative Hemodynamic Optimization Using the NICOM Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitario La Paz (Other)
Collaborators: University Hospital of the Nuestra Señora de Candelaria (Other); Hospital del Rio Hortega (Other); Hospital General de Ciudad Real (Other); University of Valencia (Other); Carmel Medical Center (Other)
Responsible Party: David Pestaña, Hospital Universitario La Paz
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: GDT NICOM
Record Dates: First submitted 2010-10-07; First posted 2010-10-08 (Estimated); Last update posted 2012-11-20 (Estimated); Status verified 2010-09

CONDITIONS: Major Abdominal Surgery
Keywords: Hemodynamic Monitoring; Goal-Directed Therapy
MeSH Terms: interventions — Hemodynamic Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual treatment (Sham Comparator): The hemodynamic management will be performed according to the institution's standard of care, using fluids at the discretion of the anesthesiologist and the ICU specialist.
  Interventions: Other: Usual treatment
- NICOM (Active Comparator): For volume replacement, crystalloids will be used following the standard procedure according to the anesthesiologist or ICU specialist. Mean arterial pressure and cardiac index will be assessed every 5 minutes, and a volume bolus (250 mL colloid in 10 minutes) will be used to achieve a:
  * Mean arterial pressure ≥ 65 mmHg (intra and postoperatively), AND
  * Cardiac index ≥ 2.5 L/min/m2 (intra and postoperatively).
  If these cardiovascular parameters are not met after the first colloid infusion, a supplementary bolus will be added. In case of not achieving the target, additional colloid boluses and/or pharmacologic support (norepinephrine in case of persistent hypotension, dobutamine in case of low cardiac output) will be provided according to the protocol
  Interventions: Device: Hemodynamic monitoring

INTERVENTIONS:
Device: Hemodynamic monitoring — Hemodynamic monitoring based on the NICOM device
  Arms: NICOM
Other: Usual treatment — Hemodynamic monitoring based on common practice
  Arms: Usual treatment

SUMMARY:
In the last years, there is a growing interest in the improvement of prognosis and shortening of hospital length of stay in high-risk surgical patients. Several evidence-based protocols ("fast-track" surgery) have been developed and implemented in some hospitals for this purpose. Cardiovascular optimization through the so-called "goal-directed therapy" (GDT) is a key element in these protocols. Previous studies in the literature use invasive monitors to assess hemodynamics. The NICOM ™ is a non-invasive monitor validated in several clinical scenarios. The aim of the present randomized, international, multi-center, open-label clinical trial is to use a GDT protocol (including colloid boluses and vasoactive drug infusion) based on data obtained from the NICOM™ device (cardiac index and mean arterial pressure) to test the hypothesis that GDT is superior to standard practice in terms of reduction in the incidence of perioperative complications and length of hospital stay in high-risk major abdominal surgery patients (requiring ICU surveillance for, at least, 24 hours). As secondary objectives, time to first flatus, wound infection, anastomotic leaks and mortality will be analysed. All patients will be followed from the day of surgery up to hospital discharge (determined by a specialist surgeon not involved in the study) or death.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients scheduled for:
* Open colorectal surgery: hemicolectomy, pancolectomy, abdomino-perineal resection.
* Gastrectomy.
* Small bowel resection.
* Signed written informed consent.

Exclusion Criteria:

* Less than 18 years old.
* Laparoscopic procedure.
* Emergency surgery.
* Intra-abdominal infection.
* Patients not requiring ICU admission (patients should stay for at least the first day at the ICU).
* Life expectancy lower than 60 days.
* Disseminated malignancy.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2011-01; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Decrease in hospital length of stay | Three months

SECONDARY OUTCOMES:
Time to peristalsis recovery | Three weeks
  Peristalsis shall be assessed by first flatus after abdominal surgery
Incidence of wound infection | Three weeks
Incidence of anastomotic leaks | Three weeks
Any cause mortality | Three months

CONTACTS AND LOCATIONS:
Overall Officials: David Pestaña, M.D. Ph.D, Principal Investigator — Hospital Universitario La Paz
Locations (4):
- Carmel Medical Center, Haifa, Israel
- Spain (3):
  - Hospital General, Ciudad Real
  - Hospital Universitario Nuestra Señora de la Candelaria, Santa Cruz de Tenerife
  - Hospital Universitario Río Hortega, Valladolid

REFERENCES:
- [Background] Squara P, Rotcajg D, Denjean D, Estagnasie P, Brusset A. Comparison of monitoring performance of Bioreactance vs. pulse contour during lung recruitment maneuvers. Crit Care. 2009;13(4):R125. doi: 10.1186/cc7981. Epub 2009 Jul 28. PMID 19638227
- [Background] Pearse R, Dawson D, Fawcett J, Rhodes A, Grounds RM, Bennett ED. Early goal-directed therapy after major surgery reduces complications and duration of hospital stay. A randomised, controlled trial [ISRCTN38797445]. Crit Care. 2005;9(6):R687-93. doi: 10.1186/cc3887. Epub 2005 Nov 8. PMID 16356219
- [Background] Lopes MR, Oliveira MA, Pereira VO, Lemos IP, Auler JO Jr, Michard F. Goal-directed fluid management based on pulse pressure variation monitoring during high-risk surgery: a pilot randomized controlled trial. Crit Care. 2007;11(5):R100. doi: 10.1186/cc6117. PMID 17822565
- [Background] Benes J, Chytra I, Altmann P, Hluchy M, Kasal E, Svitak R, Pradl R, Stepan M. Intraoperative fluid optimization using stroke volume variation in high risk surgical patients: results of prospective randomized study. Crit Care. 2010;14(3):R118. doi: 10.1186/cc9070. Epub 2010 Jun 16. PMID 20553586
- [Background] Gan TJ, Soppitt A, Maroof M, el-Moalem H, Robertson KM, Moretti E, Dwane P, Glass PS. Goal-directed intraoperative fluid administration reduces length of hospital stay after major surgery. Anesthesiology. 2002 Oct;97(4):820-6. doi: 10.1097/00000542-200210000-00012. PMID 12357146